CLINICAL TRIAL: NCT00947921
Title: POP Study: Plasty or Prosthesis to Treat Functional Mitral Regurgitation in Low Ejection Fraction Patients; a Randomized Prospective Controlled Study
Brief Title: Plasty or Prosthesis to Treat Functional Mitral Regurgitation
Acronym: POP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiochirurgia E.H. (Other)
Responsible Party: Principal Investigator, Luca Weltert, Project Leader Luca Weltert, Cardiochirurgia E.H.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00-01
Record Dates: First submitted 2009-07-23; First posted 2009-07-28 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Functional Mitral Regurgitation
Keywords: Functional MItral regurgitation
MeSH Terms: interventions — Prostheses and Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plasty (Active Comparator): Patients treated with restrictive Annuloplasty
  Interventions: Procedure: Plasty
- Prosthesis (Active Comparator): Patients treated with valve replacement
  Interventions: Procedure: Prosthesis

INTERVENTIONS:
Procedure: Plasty — Restrictive Annuloplasty
  Arms: Plasty
Procedure: Prosthesis — Valve replacement
  Arms: Prosthesis

SUMMARY:
Functional Mitral regurgitation is a now well known entity due to tethering of the valve either mono-lateral, as happens in lateral myocardial infarction, or bilateral as happens in dilated cardiomyopathy. Treatment of this pathology, either conserving the valve and addressing regurgitation by mean of restrictive annuloplasty, or implanting a prosthesis remains controversial in terms of mid and long term benefit for the patient. The investigators propose a randomized controlled study to compare the efficacy of both technique in terms of mortality and freedom from reintervention.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting for surgery due to functional mitral regurgitation

Exclusion Criteria:

* Associated Heart Surgery procedures other than CABG, Tricuspid Regurgitation correction, Atrial Fibrillation Correction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-08; Primary Completion 2016-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Mortality | 1 year of follow up after discharge from hospital

SECONDARY OUTCOMES:
Freedom from reintervention | 1 year of follow-up after discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Luca Weltert, MD, Principal Investigator — Cardiochirurgia E.H.
Locations (1):
- Divisione di Cardiochirurgia, E.H., Rome, Italy